CLINICAL TRIAL: NCT04338919
Title: A Prospective, Randomised, Open-labeled, Parallel Group Study to Assess the Effect of Optimized Antiplatelet Therapy on the Prognosis of ACS Patients With Non-predominant Coronary Artery Disease After PCI
Brief Title: Optimized Antiplatelet Therapy on the Prognosis of ACS Patients With Non-predominant Coronary Artery Disease After PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Lianglong Chen, Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optimized-APT
Record Dates: First submitted 2020-03-28; First posted 2020-04-08 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: antiplatelet therapy; Non-predominant coronary artery disease; Ticagrelor; aspirin
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention; Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O-APT group (Experimental): Ticagrelor 90 mg twice daily plus aspirin 100mg once daily in the first month, Ticagrelor 90mg bid between the second and the sixth months Ticagrelor 45mg bid between the seventh and the twelfth months
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Ticagrelor plus aspirin
- S-APT group (Active Comparator): ticagrelor 90 mg twice daily plus aspirin 100mg once daily for 12 months
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Ticagrelor plus aspirin

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — PCI with stent implantation
  Other Names: PCI
Drug: Ticagrelor plus aspirin — Ticagrelor plus aspirin

SUMMARY:
The study is to evaluate the effect of optimized 12-month step-down antiplatelet therapy (APT) compared with standard 12-month dual antiplatelet therapy in clinical net adverse events, cardiovascular and cerebrovascular adverse events and reducing clinical related bleeding events in the patients with acute coronary syndrome (ACS) who are not the predominant coronary artery disease after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is a prospective, multi- center, randomized, parallel-group trial designed to evaluate the effect of optimized 12-month step-down antiplatelet therapy compared with standard 12-month dual antiplatelet therapy in clinical net adverse clinical events, cardiovascular and cerebrovascular adverse events and reducing clinical related bleeding events in the patients with acute coronary syndrome who are not the main coronary artery disease.2020 subjects will be enrolled. After PCI,eligible patients will be randomly assigned in a 1:1 ratio to either the optimized antiplatelet therapy group（O-APT）or the standard antiplatelet therapy group（S-APT）. The primary efficacy end points are clinical net adverse clinical events ,or the event rate of the composite of cardiovascular death, non-fatal myocardial infarction, stent thrombosis, ischemia driven coronary revascularization and stroke at 12 months. The primary safety end point is the incidence of PLATO major bleeding or Bleeding Academic Research Consortium (BARC) type 2, 3 or 5 bleeding at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients admission for coronary artery disease treatment with non-emergency percutaneous intervention with stent deployment
* Enrollment into the study will require meeting at least one of these clinical syndromes.

  1. Unstable angina
  2. Non-ST elevation myocardial infarction (NSTEMI)
  3. ST elevation MI (STEMI)
* Non predominant coronary artery disease, it is defined as: exclusion of left main artery disease or left main artery bifurcated disease or ostial left anterior descending disease by coronary angiography imaging, and other high-risk vascular diseases considered by surgeons
* Patients understands the study requirements and the treatment procedures and provided informed consent before the procedure

Exclusion Criteria:

* Complications during stenting for coronary artery disease
* Stroke within 3 months or any permanent neurologic deficit, and prior intracranial bleed, or any intracranial disease such as aneurysm or fistula
* Any planned surgery within 6 months
* any reason why any antiplatelet therapy might need to be discontinued within 12 months
* Severe chronic kidney disease defined as an estimated glomerular filtration rate (eGFR) < 15ml/min/1.73m^2
* Need for chronic oral anticoagulation (warfarin/coumadin or direct oral anticoagulants)
* Platelet count < 100,000 mm^3
* Contraindication to aspirin
* Contraindication to ticagrelor
* Liver cirrhosis
* Women of child-bearing potential
* Life expectancy < 1 year
* Any condition likely to interfere with study processes including medication compliance or follow-up visits (e.g. dementia, alcohol abuse, severe frailty, long distance to travel for follow-up visits, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2020 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular and cerebrovascular adverse events | Up to 12 months after PCI
  Participants with death from cardiovascular causes, non-fatal myocardial infarction, stent thrombosis,Ischemia driven coronary revascularization and ischemic stroke.Intention to treat (ITT) analysis of whole population. Events were adjudicated by an endpoint committee.
Major bleeding events | Up to 12 months after PCI
  Plato massive hemorrhage events, including fatal hemorrhage, intracranial hemorrhage, pericardial hemorrhage with pericardial tamponade, hypovolemic shock or severe hypotension caused by hemorrhage, requiring pressor or surgery, hemoglobin level dropping 5.0 g or more per deciliter, or at least requiring blood transfusion. Events were adjudicated by an endpoint committee.
  BARC type 2, 3 or 5 bleeding. Events were adjudicated by an endpoint committee.
The net adverse clinical events | Up to 12 months after PCI
  included major adverse cardiovascular and cerebrovascular events or major bleeding events.

SECONDARY OUTCOMES:
Participants with myocardial infarction (MI) event. | Up to 36 months after PCI
  Number of participants with MI event. Events were adjudicated by an endpoint committee.
Participants with death from cardiovascular causes. | Up to 36 months after PCI
  Number of participants with death from cardiovascular causes. Events were adjudicated by an endpoint committee.
Participants with death from any cause. | Up to 36 months after PCI
  Number of participants with death from any cause. Events were adjudicated by an endpoint committee.
PLATO-defined any bleeding event. | Up to 36 months after PCI
  Number of participants with any other bleeding events (minor bleeding or minimal bleeding) as defined by the PLATO. Events were adjudicated by an endpoint committee.

OTHER OUTCOMES:
PLATO-defined any minor bleeding event | Up to 36 months after PCI
  To compare two intensities of ticagrelor therapy on minor bleeding event as any bleeding requiring medical intervention but not meeting the criteria for major bleeding. Events were adjudicated by an endpoint committee.
PLATO-defined any minimal bleeding event | Up to 36 months after PCI
  To compare two intensities of ticagrelor therapy on minimal bleeding event as all other bleeding(eg, bruising, bleeding gums, oozing from injection site) not requiring intervention or treatment.Events were adjudicated by an endpoint committee.
Other adverse events | Up to 36 months after PCI
  To compare two intensities of ticagrelor therapy on other adverse events including dyspnea or bradyarrhythmia. Events were adjudicated by an endpoint committee.
Increase of serum uric acid or creatinine | Up to 36 months after PCI
  To compare two intensities of ticagrelor therapy on increase of serum uric acid or creatinine.Events were adjudicated by an endpoint committee.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lianglong, MD, PhD, Principal Investigator — Fujian Medical University
Locations (1):
- Department of Cardiology, Union Hospital, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No